CLINICAL TRIAL: NCT05155306
Title: Relative Bioavailability of Two Different Tablet Formulations of BI 1358894 Administered in Healthy Subjects in Fasted and Fed State (an Open-label, Randomised, Single-dose, Four-period, Four-sequence Crossover Study)
Brief Title: A Study in Healthy People to Compare 2 Different Formulations of BI 1358894 Tablets Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0020; 2021-004880-28 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2021-12-13 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 1358894 - test - fasted (Experimental): A single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning following an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1358894, intended Commercial Formulation (iCF) (T)
- BI 1358894 - test - fed (Experimental): A single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning following a high-fat, high-calorie meal.
  Interventions: Drug: BI 1358894, intended Commercial Formulation (iCF) (T)
- BI 1358894 - reference - fasted (Experimental): A single dose of 100 mg (milligram) BI 1358894 given orally as two 50 mg film-coated tablets in the morning following an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1358894, Trial Formulation 2 (TFII) (R)
- BI 1358894 - reference - fed (Experimental): A single dose of 00 mg (milligram) BI 1358894 given orally as two 50 mg film-coated tablets in the morning following a high-fat, high-calorie meal.
  Interventions: Drug: BI 1358894, Trial Formulation 2 (TFII) (R)

INTERVENTIONS:
Drug: BI 1358894, intended Commercial Formulation (iCF) (T) — A single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning
  Arms: BI 1358894 - test - fasted; BI 1358894 - test - fed
Drug: BI 1358894, Trial Formulation 2 (TFII) (R) — A single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning.
  Arms: BI 1358894 - reference - fasted; BI 1358894 - reference - fed

SUMMARY:
To investigate the relative bioavailability of the intended Commercial Formulation (iCF) (Test, T) compared with Trial Formulation 2 (TFII) (Reference, R) and to assess potential food effects following oral administration of BI 1358894.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subject, or female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus one additional barrier
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus one additional barrier
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS), plus one additional barrier
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant plus one additional barrier
  * Bilateral tubal ligation plus one additional barrier
  * Surgically sterilised (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, open-label, single-dose, four-period and four-sequence crossover trial in healthy male and female subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Test Fasted - Reference Fasted - Test Fed - Reference Fed: Four-period crossover with Reference and Test treatments given under either fed or faster condition in the following order: Test fasted - Reference fasted - Test fed - Reference fed, treatments were separated by a wash-out phase of at least 17 days.
  Reference: a single dose of 100 mg (milligram) BI 1358894 given orally as of two 50 mg film-coated tablets in the morning.
  Test: a single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning.
  Fed: treatment given following a high-fat, high-calorie meal.
  Fasted: treatment following an overnight fast of at least 10 hours.
- Reference Fasted - Test Fasted - Reference Fed - Test Fed: Four-period crossover with Reference and Test treatments given under either fed or faster condition in the following order: Reference fasted - Test fasted - Reference fed - Test fed, treatments were separated by a wash-out phase of at least 17 days.
  Reference: a single dose of 100 mg (milligram) BI 1358894 given orally as of two 50 mg film-coated tablets in the morning.
  Test: a single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning.
  Fed: treatment given following a high-fat, high-calorie meal.
  Fasted: treatment following an overnight fast of at least 10 hours.
- Test Fed - Reference Fed - Reference Fasted - Test Fasted: Four-period crossover with Reference and Test treatments given under either fed or faster condition in the following order: Test fed - Reference fed - Reference fasted - Test fasted, treatments were separated by a wash-out phase of at least 17 days.
  Reference: a single dose of 100 mg (milligram) BI 1358894 given orally as of two 50 mg film-coated tablets in the morning.
  Test: a single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning.
  Fed: treatment given following a high-fat, high-calorie meal.
  Fasted: treatment following an overnight fast of at least 10 hours.
- Reference Fed - Test Fed - Test Fasted - Reference Fasted: Four-period crossover with Reference and Test treatments given under either fed or faster condition in the following order: Reference fed - Test fed - Test fasted - Reference fasted, treatments were separated by a wash-out phase of at least 17 days.
  Reference: a single dose of 100 mg (milligram) BI 1358894 given orally as of two 50 mg film-coated tablets in the morning.
  Test: a single dose of 100 mg (milligram) BI 1358894 given orally as a film-coated tablet in the morning.
  Fed: treatment given following a high-fat, high-calorie meal.
  Fasted: treatment following an overnight fast of at least 10 hours.
Period: Period 1
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out Period 1 to 2
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Period: Period 2
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 4
Completed | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out Period 2 to 3
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 4
Completed | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 4
Completed | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out Period 3 to 4
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 6 | 6 | 6 | 4
Completed | 3 | 5 | 5 | 3
Not Completed | 3 | 1 | 1 | 1
Not completed — Temporal availability | 3 | 1 | 1 | 1
Period: Period 4
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted
Started | 3 | 5 | 5 | 3
Completed | 3 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All subjects who were treated with at least one dose of the trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Fasted - Reference Fasted - Test Fed - Reference Fed | Reference Fasted - Test Fasted - Reference Fed - Test Fed | Test Fed - Reference Fed - Reference Fasted - Test Fasted | Reference Fed - Test Fed - Test Fasted - Reference Fasted | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (6.5) | 36.2 (7.5) | 44.5 (13.0) | 34.2 (6.0) | 39.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 3 | 8
  Male | 5 | 3 | 5 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 34, 48, 72, 96, 120, 144, 240 and 312 hours following drug administration in each treatment period.
Population: All subjects who were treated with at least one dose of the trial drug and who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability were included in the pharmacokinetic analysis set (PKS). Only subjects with non-missing results were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/Liter
Groups:
- BI 1358894 - Reference - Fed: A single dose of 100 mg (milligram) BI 1358894 given orally as two 50 mg film-coated tablets in the morning following a high-fat, high-calorie meal.
Arm/Group | BI 1358894 - Test - Fasted | BI 1358894 - Test - Fed | BI 1358894 - Reference - Fasted | BI 1358894 - Reference - Fed
Number analyzed (Participants) | 21 | 21 | 21 | 20
hours*nanomole/Liter | 7360 (38.7) | 14700 (26.3) | 8430 (28.6) | 14900 (26.6)
Statistical Analysis 1: Comparison: BI 1358894 - Test - Fasted vs BI 1358894 - Reference - Fasted; Analysis of variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; Geometric mean ratio [%] = 89.1, 90% CI 2-sided [79.5 to 99.7] — Ratio is calculated as test/reference. Geometric Standard Error = 1.067
Statistical Analysis 2: Comparison: BI 1358894 - Test - Fed vs BI 1358894 - Reference - Fed; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 98.1, 90% CI 2-sided [94.4 to 101.9] — Ratio is calculated as test/reference. Geometric Standard Error = 1.022
Statistical Analysis 3: Comparison: BI 1358894 - Test - Fasted vs BI 1358894 - Test - Fed; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 202.4, 90% CI 2-sided [180.1 to 227.5] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.069
Statistical Analysis 4: Comparison: BI 1358894 - Reference - Fasted vs BI 1358894 - Reference - Fed; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 173.8, 90% CI 2-sided [158.3 to 190.8] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.055

2. Primary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1358894 in plasma (Cmax).
Time Frame: as for outcome 1
Population: All subjects who were treated with at least one dose of the trial drug and who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability were included in the pharmacokinetic analysis set (PKS).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Groups:
- BI 1358894 - Fasted - Test: 100 mg (milligram) BI 1358894 given orally as a film-coated tablet once a day in the morning following an overnight fast of at least 10 hours.
- BI 1358894 - Fed - Test: 100 mg (milligram) BI 1358894 given orally as a film-coated tablet once a day in the morning following a high-fat, high-calorie meal.
- BI 1358894 - Fasted - Reference: 100 mg (milligram) BI 1358894 given orally as two 50 mg film-coated tablet once a day in the morning following an overnight fast of at least 10 hours.
- BI 1358894 - Fed - Reference: 100 mg (milligram) BI 1358894 given orally as two 50 mg film-coated tablet once a day in the morning following a high-fat, high-calorie meal.
Arm/Group | BI 1358894 - Fasted - Test | BI 1358894 - Fed - Test | BI 1358894 - Fasted - Reference | BI 1358894 - Fed - Reference
Number analyzed (Participants) | 21 | 21 | 21 | 21
nanomole/Liter | 292 (54.9) | 445 (26.1) | 378 (52.3) | 440 (23.2)
Statistical Analysis 1: Comparison: BI 1358894 - Fasted - Test vs BI 1358894 - Fasted - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 83.0, 90% CI 2-sided [69.6 to 99.0] — Ratio is calculated as test/reference. Geometric Standard Error = 1.106
Statistical Analysis 2: Comparison: BI 1358894 - Fed - Test vs BI 1358894 - Fed - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 99.7, 90% CI 2-sided [88.7 to 112.0] — Ratio is calculated as test/reference. Geometric Standard Error = 1.070
Statistical Analysis 3: Comparison: BI 1358894 - Fasted - Test vs BI 1358894 - Fed - Test; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 153.6, 90% CI 2-sided [126.0 to 187.3] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.121
Statistical Analysis 4: Comparison: BI 1358894 - Fasted - Reference vs BI 1358894 - Fed - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 121.4, 90% CI 2-sided [99.6 to 147.8] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.120

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/Liter
Arm/Group | BI 1358894 - Fasted - Test | BI 1358894 - Fed - Test | BI 1358894 - Fasted - Reference | BI 1358894 - Fed - Reference
Number analyzed (Participants) | 21 | 21 | 21 | 20
hours*nanomole/Liter | 8020 (37.3) | 16100 (30.3) | 9120 (28.0) | 15900 (28.1)
Statistical Analysis 1: Comparison: BI 1358894 - Fasted - Test vs BI 1358894 - Fasted - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 89.9, 90% CI 2-sided [80.4 to 100.4] — Ratio is calculated as test/reference. Geometric Standard Error = 1.066
Statistical Analysis 2: Comparison: BI 1358894 - Fed - Test vs BI 1358894 - Fed - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 100.4, 90% CI 2-sided [96.8 to 104.1] — Ratio is calculated as test/reference. Geometric Standard Error = 1.021
Statistical Analysis 3: Comparison: BI 1358894 - Fasted - Test vs BI 1358894 - Fed - Test; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 202.6, 90% CI 2-sided [179.6 to 228.5] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.072
Statistical Analysis 4: Comparison: BI 1358894 - Fasted - Reference vs BI 1358894 - Fed - Reference; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio [%] = 172.3, 90% CI 2-sided [158.2 to 187.7] — Ratio is calculated as fed/fasted. Geometric Standard Error = 1.050

ADVERSE EVENTS:
Time Frame: All-cause Mortality: from time of administration till the end of study (EoS) examination, time of next administration or trial termination. Up to 25 days. Adverse events: from time of administration till the end of the residual effect period, time of next administration or trial termination, whichever occurs first. Up to 17 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Arm/Group | BI 1358894 - Reference - Fasted | BI 1358894 - Reference - Fed | BI 1358894 - Test - Fasted | BI 1358894 - Test - Fed
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 15/21 | 13/21 | 13/21 | 13/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1358894 - Reference - Fasted (N=21) | BI 1358894 - Reference - Fed (N=21) | BI 1358894 - Test - Fasted (N=21) | BI 1358894 - Test - Fed (N=21)
Headache (Nervous system disorders) | 14 | 13 | 12 | 10
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0
COVID-19 (Infections and infestations) | 3 | 1 | 1 | 3
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05155306/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT05155306/SAP_001.pdf